CLINICAL TRIAL: NCT05004051
Title: Prospective Registry Study to Collect Imaging and Clinical Data on Patients With Aortic Aneurysm Disease Undergoing Serial Monitoring & Pre and Post Endovascular Repair
Brief Title: ViTAA Registry Pre- and Post-Operative Monitoring for Endovascular Aortic Aneurysm Repair and Serial Monitoring for AAA
Status: Recruiting | Type: Observational
Sponsor: ViTAA Medical Solutions (Industry)
Responsible Party: Principal Investigator, Dr Mark Farber, Principal Investigator, ViTAA Medical Solutions
Other Study IDs: CIP-ViTAA-001
Record Dates: First submitted 2021-07-29; First posted 2021-08-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Abdominal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Patients who are booked for and then subsequently have undergone endovascular repair.: Patients who are scheduled and ultimately receive on-IFU endovascular infrarenal aortic aneurysm repair (EVAR)
  Interventions: Device: ViTAA Analysis
- Patients with infrarenal AA without indications for repair undergoing serial monitoring: Patients who do not yet qualify for the aortic aneurysm repair who are enrolled in a serial monitoring program
  Interventions: Device: ViTAA Analysis

INTERVENTIONS:
Device: ViTAA Analysis — Imaging Analysis Software

SUMMARY:
This is a Prospective Registry study to collect imaging and clinical data both on patients with aortic aneurysm disease undergoing serial monitoring and on patients pre and post-endovascular repair, using ViTAA (The Sponsor) aortic mapping technology.

DETAILED DESCRIPTION:
This a prospective, multi-center, registry of patients that are being assessed with the ViTAA software. Patients will be enrolled at selected North American centers in the US and Canada. The Registry will enroll patients from the following two populations:

* patients who are scheduled and ultimately receive endovascular infrarenal aortic aneurysm repair (EVAR);
* patients who do not yet qualify for infrarenal aortic aneurysm repair based on anatomic size criteria who are enrolled in a serial monitoring program.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged 18 years or over
2. Infrarenal Aortic Aneurysm ≥ 45 mm in diameter.
3. Patient meets on-IFU criteria for endovascular reconstruction

Exclusion Criteria:

1. Patient has a known or clinically suspected major connective tissue disorder, autoimmune disorder, vasculitis, or aortic dissection.
2. Patient has renal failure (defined as dialysis dependent or serum creatinine ≥2.0mg/dL or 175umol/L
3. Patients with previous aortic reconstruction in the involved segment.
4. Patients receiving oral or parenteral corticosteroid therapy for other unrelated disease. (Excludes inhaled corticosteroids).
5. Patient has a sensitivity to contrast imaging agents.
6. Patient has aortic dissection.
7. Patient has atrial fibrillation.
8. Patient has arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients who are booked for and then subsequently have undergone endovascular repair.
  2. Patients with infrarenal aortic aneurysms without indications for repair undergoing serial monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of aneurysm rupture or critical growth. | 6 months
  * Critical growth defined as an increase of > 0.5 cm in any of the three growth measurements below
  * Critical growth defined as an increase of > 0.5 cm in aortic diameter.
  * Critical growth defined as an increase of > 0.5 cm in ILT.
  * Critical growth defined as an increase of > 0.5 cm in aneurysm sac volume.
Composite of aneurysm rupture or critical growth. | 1 year
  * Critical growth defined as an increase of > 0.5 cm in any of the three growth measurements below
  * Critical growth defined as an increase of > 0.5 cm in aortic diameter.
  * Critical growth defined as an increase of > 0.5 cm in ILT.
  * Critical growth defined as an increase of > 0.5 cm in aneurysm sac volume.

SECONDARY OUTCOMES:
CHUM Ancillary Ultrasound Study | 6 months
  For patients recruited at the CHUM:
  1. Correlation between ultrasound and multiphase CT based strain and RAW values
  2. Correlation between AAA growth and ultrasound-based strain and RAW maps
CHUM Ancillary Ultrasound Study | 1 year
  For patients recruited at the CHUM:
  1. Correlation between ultrasound and multiphase CT based strain and RAW values
  2. Correlation between AAA growth and ultrasound-based strain and RAW maps

CONTACTS AND LOCATIONS:
Overall Officials: Mark Farber, Principal Investigator — University of North Carolina, Chapel Hill
Locations (8):
- United States (4):
  - UAB - University of Alabama in Birmingham Hospital, Birmingham, Alabama
  - MGH - Massachusetts General Hospital Fireman Vascular Center, Boston, Massachusetts
  - UNC - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Washington, Seattle, Washington
- Canada (4):
  - UCGY - University of Calgary, Peter Lougheed Center, Calgary, Alberta
  - UHN - University Health Network - Toronto General Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - MUHC - McGill University Health Centre, Montreal, Quebec